CLINICAL TRIAL: NCT02381886
Title: A Phase I Study of IDH305 in Patients With Advanced Malignancies That Harbor IDH1R132 Mutations
Brief Title: A Study of IDH305 in Patients With Advanced Malignancies That Harbor IDH1R132 Mutations
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIDH305X2101
Record Dates: First submitted 2015-03-02; First posted 2015-03-06 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Advanced Malignancies That Harbor IDHR132 Mutations
Keywords: IDHR132 mutations; IDH305; IDH; IDH1; AML; Acute Myeloid Leukemia; Leukemia; Myeloid; Acute; MDS; Myelodysplastic Syndrome; Glioma; Oligodendroglioma; Astrocytoma; Glioblastoma; Cholangiocarcinoma; Solid Tumors
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia; Myelodysplastic Syndromes; Glioma; Oligodendroglioma; Astrocytoma; Glioblastoma; Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IDH305 (Experimental)
  Interventions: Drug: IDH305

INTERVENTIONS:
Drug: IDH305

SUMMARY:
A Phase I study of IDH305 in patients with advanced malignancies that harbor IDH1R132 mutations.

ELIGIBILITY:
Inclusion Criteria:

* Documented IDH1R132-mutant tumors
* ECOG performance status ≤ 2

Exclusion Criteria:

* Patients who have received prior treatment with a mutant-specific IDH1 inhibitor (with the exception of glioma patients)
* Medical conditions that would prevent the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures such as the presence of other clinically significant cardiac, respiratory, gastrointestinal, renal, hepatic or neurological disease.
* Acute Promyelocytic Leukemia
* Women who are pregnant or lactating

Other protocol-defined Inclusion/Exclusion may apply

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2015-03-06 (Actual); Primary Completion 2016-12-07 (Actual); Study Completion 2027-02-10 (Estimated)

PRIMARY OUTCOMES:
Incident rate of dose limiting toxicities (DLTs) | 21 days
  To estimate the maximum tolerated dose/recommended dose for expansion (MTD/RDE)

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | 30 months
  To characterize the safety and tolerability of IDH305
Plasma PK parameters (AUC, Cmax, Tmax) | 30 months
  To characterize the PK profile of IDH305
Changes of 2-hydroxyglutarate concentration in patient specimens | 30 months
  To characterize the PD profile of IDH305
Overall response rate (ORR) | 30 months
  To assess any preliminary anti-tumor activity of IDH305
Incidence of serious adverse events (SAE) | 30 months
  To characterize the safety and tolerability of IDH305

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (16):
- United States (5):
  - Dana Farber Cancer Institute SC (1), Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Columbia University Medical Center- New York Presbyterian Onc Dept., New York, New York
  - Columbia University Medical Center, New York, New York
  - Uni Of TX MD Anderson Cancer Cntr, Houston, Texas
- Australia (2):
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Parkville, Victoria
- Novartis Investigative Site, Leuven, Belgium
- Novartis Investigative Site, Toronto, Ontario, Canada
- Germany (3):
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Heidelberg
- Netherlands (2):
  - Novartis Investigative Site, Rotterdam, South Holland
  - ErasmusMC Cancer lnstitute, Neuro-Oncology, Rm G3-55, Rotterdam
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] DiNardo CD, Hochhaus A, Frattini MG, Yee K, Zander T, Kramer A, Chen X, Ji Y, Parikh NS, Choi J, Wei AH. A phase 1 study of IDH305 in patients with IDH1R132-mutant acute myeloid leukemia or myelodysplastic syndrome. J Cancer Res Clin Oncol. 2023 Mar;149(3):1145-1158. doi: 10.1007/s00432-022-03983-6. Epub 2022 Mar 30. PMID 35353219